CLINICAL TRIAL: NCT01385618
Title: Analysis of Gene-polymorphisms Relating to Human Subfertility: Estradiol-receptor-polymorphism and Progesterone-receptor-polymorphism
Brief Title: Gene-polymorphisms Relating to Human Subfertility
Status: Completed | Type: Observational
Sponsor: Infertility Treatment Center Dortmund (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Dieterle, Prof. Dr., Infertility Treatment Center Dortmund
Other Study IDs: PRP-ERP2010
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Estradiol Receptor Polymorphism; Progesterone Receptor Polymorphism; IVF; Subfertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- high responder: females with >15 follicles or E2>3000 after treatment with gonadotropins
- low responder: patients with <3 follicles or no response to treatment with gonadotropins
- control: females with an indication for treatment because of male subfertility

SUMMARY:
Estradiol is synthesized by granulosa cells of ovaries under control of follicle-stimulating hormone (FSH) and luteinizing hormone (LH). It is known that Estradiol plays a crucial role in maturation and fertilization of oocytes. Furthermore it is involved in development of secondary female sexual organs, fertility and maintenance of pregnancy.

Estradiol influences these processes by binding to estradiol receptors (ER). They are ligand-depending transcription-factors. In humans there are two subtypes: ERa and ERb, which are synthetized from gene ESR1 on chromosome 6 and ESR2 on chromosome 14. Both subtypes are expressed in the ovary. Both genes are polymorph. Especially for ERa subtype several polymorphisms and mutations are known which can be linked to breast cancer, spontaneous abortions, osteoporosis and the point in time of menarche. Furthermore some studies have shown a relationship between certain polymorphisms and the risk of infertility associated gynecological malfunctions and the result of IVF treatments.

Progesterone is a hormone which plays a crucial role in initiation and maintenance of pregnancy. It induces the transformation of the endometrium, which facilitates the implantation of the fertilized oocyte and supports the pregnancy. Progesterone acts by binding to its receptor. The gene for this receptor is polymorph within the population, whereas some variants seem to account for implantation failure of embryos.

In the investigators study the investigators will analyse the role of ERP and PRP polymorphisms in the context of IVF treatment. The analyzed genotypes are two polymorphisms of ESRI, called Pvu and Xba, as well as a variant of ESRII, ER2. In the progesterone receptor gene a single nucleotide exchange at position +331 (G->A) plays a role.

The parameters correlated with are concentrations of estradiol, progesterone and FSH, number of follicles, number of fertilized oocytes and pregnancy rate.

The investigators hope to optimize established treatment protocols and to improve the chances of success of IVF treatments depending on the genotype of the patient.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ ICSI treatment with hormonal stimulation
* reproductive age
* high response OR low response OR male subfertility

Exclusion Criteria:

* other fertility treatments like IUI or timed intercourse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients at reproductive age seeking IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
genetic testing for two estrogene receptor genes, correlating to numbers of oocytes retrieved at oocyte punction after hormonal stimulation | 30.06.2013

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Neuer, Principal Investigator — Infertility Treatment Center Dortmund
Locations (1):
- Infertility treatment center Dortmund, Dortmund, North Rhine-Westphalia, Germany